CLINICAL TRIAL: NCT05539209
Title: OKquit -- Testing a Novel Smartphone Application for Smoking Cessation With the Oklahoma Helpline
Brief Title: Testing a Novel Smartphone Application for Smoking Cessation With the Oklahoma Helpline
Acronym: OKquit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14792
Record Dates: First submitted 2022-09-06; First posted 2022-09-14 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Standard Helpline Care (SC) group (Active Comparator): The SC group will receive standard Oklahoma Smoking Cessation Helpline care AND complete daily check-ins and weekly surveys for 27 weeks.
  Interventions: Behavioral: Standard Helpline Care
- OKquit group (Active Comparator): The OKquit group will receive SC plus daily check-ins and weekly surveys for 27 weeks. In addition, the OKquit group will receive tailored smoking cessation messages in the smartphone application following completion of each survey. Further, the OKquit group will have access to on-demand smoking cessation content through the app.
  Interventions: Behavioral: OKquit

INTERVENTIONS:
Behavioral: OKquit — Standard Oklahoma Helpline care plus smartphone-based daily check-ins and weekly surveys plus OKquit Smartphone App including tailored messages and on-demand content designed to assist participants in their cessation attempt.
  Arms: OKquit group
Behavioral: Standard Helpline Care — Standard Oklahoma Helpline care plus smartphone-based daily check-ins and weekly surveys.
  Arms: The Standard Helpline Care (SC) group

SUMMARY:
Over 470,000 tobacco users have been served by the Oklahoma Tobacco Helpline (OTH). The OTH reaches a substantial number of smokers each year, but follow-up rates are notoriously low and many smokers may prefer smartphone-based smoking cessation interventions rather than web- or phone-based OTH programming (e.g., counseling). Highly flexible and low burden technology-based treatment approaches may overcome barriers that have limited the use and effectiveness of traditional smoking cessation treatments among underserved adult smokers (e.g., racial/ethnic minorities, rural residence, low socioeconomic status). This study is a randomized controlled trial that will evaluate the feasibility and initial efficacy of an innovative, evidence-based smoking cessation app tailored for smokers that contact the OTH for services. A total of 500 treatment-seeking men and women will be randomly assigned to receive either Standard Helpline Care plus brief (30 second) daily check-ins and weekly smartphone-based surveys through the Insight app (SC) or SC plus the OKquit smoking cessation app (OKq). All participants will receive standard Helpline services (e.g., nicotine replacement therapy), but only the OKq group will receive on-demand content and tailored messages through the app. All participants will be followed for 27 weeks after they are randomized to an intervention group and complete smartphone-based survey assessments. Participants that report smoking abstinence during the 26-week EMA will be sent a low-cost carbon monoxide monitor to verify smoking status.

DETAILED DESCRIPTION:
Over 470,000 tobacco users have been served by the Oklahoma Tobacco Helpline (OTH). The OTH reaches a substantial number of smokers each year, but follow-up rates are notoriously low and many smokers may prefer smartphone-based smoking cessation interventions rather than web- or phone-based OTH programming (e.g., counseling). Highly flexible and low burden technology-based treatment approaches may overcome barriers that have limited the use and effectiveness of traditional smoking cessation treatments among underserved adult smokers (e.g., racial/ethnic minorities, rural residence, low socioeconomic status). This study is a randomized controlled trial that will evaluate the feasibility and initial efficacy of an innovative, evidence-based smoking cessation app tailored for smokers that contact the OTH for services. A total of 500 treatment-seeking men and women will be randomly assigned to receive either Standard Helpline Care plus brief (30 second) daily check-ins and weekly smartphone-based surveys through the Insight app (SC) or SC plus the OKquit smoking cessation app (OKq). All participants will receive standard Helpline services (e.g., nicotine replacement therapy), but only the OKq group will receive on-demand content and tailored messages through the app. All participants will be followed for 27 weeks after they are randomized to an intervention group and complete smartphone-based survey assessments. Participants that report smoking abstinence during the 26-week EMA will be sent a low-cost carbon monoxide monitor to verify smoking status.

PROPOSED PROCEDURE:

Individuals who call the OTH will be asked if they own a smartphone (>85% of US adults currently own a smartphone). Those that own a smartphone that is compatible with our Insight™ mHealth Platform will be asked if they are interested in participating in this study. Interested individuals will be sent a link to the REDCap study screener by phone, email, or text (via OTH provider and/or this research team) so that they can complete the study screener. Those that qualify for the study will be called by Dr. Businelle's research team to complete informed consent, finalize enrollment, and be randomized into a study group. All participants will use a version of the Insight™ app (i.e., SC assessment only app or OKquit app which contains assessments and intervention content) to complete a brief Baseline survey. Upon completion of the Baseline survey, participants will be randomized to an intervention group and use the app to set a quit date within the next 21 days. Note: A minimization technique will be used to ensure that groups are balanced by race (white vs. non-white), biological sex (male vs. female), and cigarettes smoked per day (<20 vs. 20 or more). During the randomization call, participants will be instructed on how to complete phone-based EMAs. Participants who do not complete the baseline assessment and randomization call will be removed from the study.

After randomization, the app will prompt a brief daily check-in (e.g., 4 questions) and weekly assessments (~30 questions; both groups). During the morning check-in assessment, all participants will elect to complete 0-5 additional brief check-ins (i.e., 2 questions) that day. Responses to these check-ins are used to collect information about relapse risk and automatically TAILOR OKq intervention messages to the participant's current needs in real-time. Consistent with the Phoenix pilot, the weekly EMA will be prompted by the smartphone app on Saturdays. The phone will ring and vibrate to cue these EMAs. This EMA will ask questions about current and past week thoughts, feelings, and behaviors. All participants (both groups) that report they did not smoke in the past 7 days during the week 26 weekly survey will be mailed a low-cost carbon monoxide monitor that has been paired with the Insight™ smartphone application to verify abstinence. All contact with research staff will occur remotely - there will be no required in person visits for this study. Participants will be compensated $20 for completing the study baseline, $5 for completing each weekly study survey for 27 weeks, and $50 for completing the app-based end of study follow-up assessment. Thus, total compensation will be up to $205 plus an additional $20 for those who complete the end of study biochemical verification of smoking abstinence (only those that report abstinence at the end of the study will be asked to verify smoking abstinence).

IMPORTANCE OF KNOWLEDGE REASONABLY EXPECTED TO RESULT FROM THE RESEARCH:

Smoking is becoming increasingly concentrated among individuals with the lowest levels of income, education, and occupational status. In fact, smoking rates in the United States among people living below the poverty line is nearly twice as high as those above the poverty threshold. Highly flexible and low burden technology-based treatment approaches may overcome many of the barriers that have limited the use and effectiveness of traditional smoking cessation treatments among adults with low socioeconomic status (SES). Ecological momentary assessment (EMA), in which mobile devices are used to capture moment-to-moment experiences, allows for the measurement of phenomena in real-time within natural settings. Smartphone-based smoking cessation apps could offer easily accessible, highly tailored, and intensive interventions at a fraction of the cost of traditional smoking cessation counseling.

ELIGIBILITY:
Inclusion Criteria:

* Are ≥ 18 years of age
* Expressed interest in participating in this study by allowing the OTH provider to share their contact details with the study research team
* Valid Oklahoma residential address to mail study materials
* Score of ≥ 4 on the Rapid Estimate of Adult Literacy in Medicine-Short Form (REALM-SF)
* Willing to quit smoking within 21 days after the randomization phone call
* Currently smoke ≥ 5 cigarettes per day
* Agree to complete daily 30 second EMA check-ins and 27 weekly 3-5 minute smartphone-based surveys
* Possession of an active smartphone that is compatible with the Insight mHealth Platform
* Agree to complete the 27-week post-randomization follow-up assessment (which may include biochemical verification of smoking abstinence)
* Provide evidence that they are a current smoker (e.g., text a picture of their pack of cigarettes when requested during the screening call)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence | 27 Weeks
  Biochemically verified smoking abstinence will be assessed using a portable carbon monoxide monitor.

SECONDARY OUTCOMES:
Treatment engagement | 27 weeks
  Engagement will be assessed via counts of completed Oklahoma Helpline service calls and number of times the OKquit app content is accessed
Cessation motivation | 27 weeks
  Cessation motivation will be assessed each week via smartphone app based survey

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Businelle, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Businelle M, Becerra J, Witten C, Chen S, Kezbers K, Beebe LA, Kendzor DE. Smartphone-Based Smoking Cessation Intervention (OKquit) for Oklahoma Tobacco Helpline Users: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Aug 1;13:e56827. doi: 10.2196/56827. PMID 39088254